CLINICAL TRIAL: NCT02040441
Title: Proteomic Prediction and Renin Angiotensin Aldosterone System Inhibition Prevention Of Early Diabetic nephRopathy In TYpe 2 Diabetic Patients With Normoalbuminuria
Acronym: PRIORITY
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peter Rossing (Other)
Collaborators: Mosaiques Diagnostics GmbH (Unknown); University Medical Center Groningen (Other); University of Glasgow (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); Univerzita Karlova v Praze (Other); Geniko Nosokomeio Athinas Ippokrateio (Unknown); Institut Klinické a Experimentální Mediciny Praze (Unknown); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Klinikum St. Georg Leipzig (Unknown); Cyril and Methodius University in Skopje (Unknown); Hannover Clinical Trial Center (Unknown); European Commission (Other); Diabetes Vascular Research Foundation Hoogeveen (Unknown); University Ghent (Other); Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden (Unknown); Stichting VUMC (Unknown); Diabetologen Hessen (Unknown)
Responsible Party: Sponsor-Investigator, Peter Rossing, Professor, Chief Physician, MD, DMSc, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2012-000452-34; 2012-000452-34 (EudraCT Number)
Record Dates: First submitted 2013-12-16; First posted 2014-01-20 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Diabetic Nephropathy; Diabetic Retinopathy
Keywords: Proteomics; Diabetes; Chronic kidney disease; Diabetic nephropathy; Diabetic retinopathy; Mineralocorticoid receptor antagonists; Spironolactone; Microalbuminuria
MeSH Terms: conditions — Diabetic Nephropathies; Diabetic Retinopathy; Diabetes Mellitus; Renal Insufficiency, Chronic | interventions — Spironolactone; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Spironolactone (Active Comparator): High-risk pattern: Spironolactone 25 mg once daily + Standard care
  Interventions: Drug: Spironolactone; Drug: Standard care
- Placebo (Placebo Comparator): High-risk pattern: One placebo tablet once daily + Standard care
  Interventions: Drug: Placebo; Drug: Standard care
- Observational (Other): Low-risk pattern: Standard care
  Interventions: Drug: Standard care

INTERVENTIONS:
Drug: Spironolactone
  Arms: Spironolactone
Drug: Placebo
  Arms: Placebo
Drug: Standard care — Standard diabetes care

SUMMARY:
This is a prospective, multicenter, randomized, double blind, placebo-controlled and a prospective observational study.

This study will be conducted at 15 study centers in various European countries. 1777 participant between 18 to 75 years old with Type 2 diabetes mellitus and normoalbuminuria participate in the study. The study period is 2 - 4.5 years (excluding the 6 week screening period). Depending on the risk score of the urinary protein pattern, participants have been stratified into an observational group or an interventional group. Participants with the low risk pattern (observational group) attend visits annually after screening and baseline. Participants with the high risk pattern (interventional group) attend study visits every 13 weeks after screening and baseline.

The interventional group has been allocated into one treatment group either receiving spironolactone or placebo. A placebo is a medicine without a pharmaceutical substance. The allocation to one of the two treatment groups has been done by a random distribution procedure established before the study start.

The results of the urine sample from the Screening visit has been analysed and the urine proteomic pattern is determined to be either low- or high risk pattern and will determine the further study program.

Participants with a low-risk pattern (observational group):

During the study period, participants attend an annual project visit, were regular diabetes care is performed and three urine samples are analysed for albuminuria.

Participants with a high-risk pattern (intervention group):

Participants with a high-risk pattern have been randomized to either spironolactone treatment or placebo. The treatment is one tablet for oral use to be taken once a day for the entire study period. Four times each year (every 13th week) a study visit is conducted including examination of three urine samples for albuminuria.

This study aims to:

1. Confirm in a prospective multicenter study of normoalbuminuric type 2 DM patients that the urinary proteome test identifies patients with a high risk for development of microalbuminuria.
2. Demonstrate the clinical utility of the test by showing that aldosterone blockade in high-risk patients can reduce progression to microalbuminuria in comparison to placebo, on the top of standard treatment in a randomized double-blind, placebo-controlled multicenter study.

DETAILED DESCRIPTION:
Background Information Diabetes mellitus (DM) affects 9% of the European population and the cost of caring for patients with DM accounts for 15% of the European health care budget expenditure. Al-most 90% of patients have type 2 DM, and absolute numbers are expected to rise in parallel to the current obesity and metabolic syndrome epidemic. Improved treatment has reduced mortality but the prolonged duration of DM increases the likelihood of development of late diabetic complications.

Diabetic nephropathy is one of the major late complications of diabetes and is associated with substantial cardiovascular morbidity and mortality and is a leading cause of end stage renal disease (ESRD) in the Western world. In clinical practice, renal impairment is diagnosed by albuminuria or proteinuria and/or changes in serum creatinine/creatinine clearance indicating alterations of the glomerular filtration rate (GFR). However, the inter-individual variability is high, and as a consequence, these standard tests have a moderate specificity and sensitivity at early stages of disease, with major limitations in the diagnosis of the early stages of diabetic nephropathy (DN).

Development of DN is generally characterized by an increase of urinary albumin excretion rate (>300 mg/24 h or 200 μg/min). Microalbuminuria (30-300 mg/24 h or 20-200 μg/min) is considered a risk factor and as an early indicator of future onset of DN. Microalbuminuria is regarded as the earliest clinical marker of renal damage. However, structural changes to the kidney have already occurred at the stage of microalbuminuria and patients with microalbuminuria have a high risk for development of renal disease, but also increased morbidity and mortality due to cardiovascular disease.

Blood pressure and glycemic control with pharmacotherapeutic intervention as well as life style interventions are the cornerstones of type 2 DM management aiming at prevention of microvascular complications. Specific therapy, particularly treatment with angiotensin converting enzyme inhibitors (ACE) and angiotensin receptor antagonists (ARB) to prevent progression to overt proteinuria and advanced stages of diabetic nephropathy is recommended if microalbuminuria is present. Studies aiming for earlier prevention of nephropathy by starting renin angiotensin aldosterone system (RAAS) blocking treatment in normoalbuminuric patients have given mixed and often disappointing results. This might reflect that a large fraction of normoalbuminuric patient may not be at risk for progression thereby reducing the event rate or power in previous studies. Early identification of normoalbuminuric patients at high risk for development of diabetic nephropathy could identify patients who might benefit of intervention with increased blockade of the RAAS. Furthermore, blockade of the RAAS with aldosterone blockade has been demonstrated to reduce urinary albumin excretion with 20-30% on top of standard antihypertensive treatment including ACE or ARB in proteinuric type 1 and 2 diabetic patients, and a 60% reduction was seen in microalbuminuric type 1 diabetic patients. Therefore, it may also hold the potential to reduce the risk of development of microalbuminuria in high risk normoalbuminuric patients.

CKD Biomarker panel Proteomics is the analysis of large number of proteins or polypeptides in tissue and body fluids. Capillary electrophoresis mass spectrometry (CE-MS) enables reproducible and robust high-resolution analysis of several thousand low-molecular-weight urinary proteins/peptides in about one hour. Urine holds several advantages over blood in clinical proteomics. It can be collected non-invasively and its proteome is relatively stable. Members of the consortium have successfully identified a urinary biomarker pattern including 273 peptides significantly associated with chronic kidney disease (CKD273).

Importantly, the biomarker panel has been validated in a multicentric approach involving >1000 blinded samples. The accuracy was high (96% sensitivity and 98% specificity), when evaluating only the diabetic patients in the test-set. To test the CKD273 pat-tern as a tool for early detection of DN, we recently performed an independent longitudinal study of normoalbuminuric diabetic patients at inclusion. The urinary CKD273 pattern distinguished progressing patients from non-progressing patients. The corresponding receiver operating characteristic (ROC) analysis resulted in an area under the curve (AUC) of 0.925 assuming a prevalence of 30% for DN. The positive predictive value was 97% and the negative predictive value was 88%. The specificity of the CKD273 pattern was further evaluated in patients without any evidence for renal impairment based on clinical history, creatinine, or urinary protein levels resulting in an overall specificity of 98%.

The used CKD273 pattern showed that these biomarkers can detect initiation and progression of DN earlier than the currently used indicators, well preceding increases in urinary albumin levels. While the CKD273 pattern detected DN with >90% accuracy four years before clinical diagnosis, serum creatinine and/or Urine albumin execration rate did not detect DN earlier than one and two years before clinical manifestation, respectively. In addition, diagnostic accuracy was significantly lower compared to the CKD273 pattern. In addition, two independent studies on type 1 and type 2 DM patients, on longitudinally collected samples over a period of 10 years demonstrate that CKD273 markers of kidney disease were altered 3 to 5 years prior to manifestation of albuminuria, and 1 to 2 years prior to development of microalbuminuria. Thus, the performance of the CKD273 pattern is better than prediction based on urinary albumin values and represents potentially a significant improvement over the current state of the art in assessing DN, enabling earlier detection with higher accuracy than urinary albumin.

Finally, the proteome analysis and application of the CKD273 pattern indicated a positive scoring for CKD in microalbuminuric type 2 diabetic patients, which showed persistent improvement during long-term renoprotective treatment with Irbesartan, while placebo treated patients showed a slight deterioration of kidney damage markers likely reflecting disease progression in the absence of preemptive intervention.

Collectively, our existing data strongly indicate that the urinary proteomics based test ap-pears ideal to identify patients who will develop microalbuminuria and ultimately DN and thereby facilitates targeting intensified preventative therapy to this group.

Rationale:

1. Urinary proteomics predicts development of microalbuminuria (as a surrogate marker for the development of overt nephropathy) in a cohort of type 2 diabetic patients with normal urinary albumin excretion at screening.
2. Early initiation of preventive therapy with spironolactone reduces risk of transition to microalbuminuria in those identified by urinary proteomics to be at high risk, and thereby delays progression to overt nephropathy. Treatment can be spared for those with low risk according to urinary proteomics, paving the way of personalised medicine

Primary Objective To confirm that urinary proteomics can predict development of microalbuminuria (as a surrogate marker for the development of overt nephropathy) in a cohort of type 2 diabetic patients with normal urinary albumin excretion.

Secondary Objectives To investigate if early initiation of preventive therapy with spironolactone 25 mg once daily reduces risk of transition to microalbuminuria in those patients identified by urinary proteomics to be at high risk.

Additional Scientific Objectives To compare the rate of change in urinary albumin excretion rate in high vs. low-risk population (based on the proteomic test), and to compare the effect of spironolactone on rate of change in urine albumin execration rate in the intervention group.

In addition, the objective is to study the rate of change in estimated GFR in relation to urinary marker pattern (CKD 273) and the intervention with spironolactone.

To study the ability of urinary proteomic patterns, to predict cardiovascular or renal events during the study as well as response to intervention, in relation to study endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be provided before participation. Patient information and consent form must be approved by relevant independent ethical committee. Specifically, all participating patients will be asked to give informed consent for long-term follow-up and collection of follow-up data
2. Male or female patients ≥ 18 years and < 75 years of age at Screening visit
3. Type 2 DM (WHO criteria)
4. Persistent normoalbuminuria (at least 2 of 3 UACR < 30 mg/g samples from "run in"-period)
5. Estimated GFR >45 ml/min/1.73m2 (MDRD formula) at Screening visit
6. The patient must be willing and able to comply with the protocol for the duration of the study
7. Female without child-bearing potential at the screening visit. Defined as one or more of following:

7.1) Female patients ≥ 50 years of age at the day of inclusion, who have been postmenopausal for at least 1 year 7.2) Female patients < 50 years of age at the day of inclusion, who have been postmenopausal for at least 1 year and serum follicle stimulating hormone levels > 40 milli International unit / mL as well as serum estrogen levels < 30 pg/ml or a negative estrogen test.

7.3) 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral ovariectomy with or without hysterectomy.

OR a negative urine pregnancy test at the Screening visit AND one or more of following:

7.4) Correct use of reliable contraception methods. This includes one or more of the following: hormonal contraceptive (such as injection, transdermal patch, implant, cervical ring or oral) or an intrauterine device (IUD) OR correct use of double barrier with one of the following: barrier methods (diaphragm, cervical cap, Lea contraceptive or condom) AND in combination with a spermicide.

7.5) General sexual abstinence from the time of screening/ baseline, during the study until a minimum of 30 days after the last administration of study medication if this is already established as the patient's preferred and usual lifestyle.

7.6) Having only female sexual partners. 7.7) Sexual relationship with sterile male partners only

Exclusion Criteria:

1. Average of systolic BP< 110 or >160 mm Hg at baseline
2. Average of diastolic BP > 100 mm Hg at baseline
3. Type 1 DM (WHO criteria)
4. HbA1c <6.5% (48 mmo l/ mol) AND > 5 years of known duration of diabetes type 2 AND never treated with an antidiabetic drug of any kind.
5. Current in treatment with more than one RAAS blocking agent (Angiotensin Converting Enzyme inhibitor, Angiotensin Receptor Blocker or Direct Renin Inhibitor)
6. Current lithium treatment
7. Known or suspected hypersensitivity to Spironolactone or to any of its excipients.
8. Current use of potassium sparing diuretics, such as: Spironolactone, Eplerenone or Amiloride etc.
9. Screening (week -6) plasma (or serum) potassium level >5.0 mmol/L
10. Low plasma sodium determine by the investigator
11. Current cancer treatment or within five years from baseline (except basal cell skin cancer or squamous cell skin cancer)
12. Any clinically significant disorder, except for conditions associated with type 2 DM history, which in the Investigators opinion could interfere with the results of the trial
13. Cardiac disease defined as: Heart failure (NYHA class III-IV) and/or diagnosis of unstable angina pectoris and/or myocardial ischemia, stroke, cardiac re-vascularisation or coronary artery bypass within the last 3 months
14. Diagnosis of non-Diabetic CKD current or in the past
15. Diagnosis of liver cirrhosis with current impaired liver function within the last 3 years.
16. Diagnosis of Addison's disease.
17. Being lactating.
18. Intend to become pregnant within the duration of the study or not use adequate birth control.
19. Known or suspected abuse of alcohol or narcotics
20. Not able to understand informed consent form
21. Participation in any other intervention trial than PRIORITY or a related sub-study is not allowed within 30 days before inclusion or concurrent to this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1777 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Albuminuria | Screening, (Low-risk: year 1, 2 and 3), (high-risk: week 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156)
  Development of confirmed microalbuminuria (UACR >30 mg/g) in at least two out of three first morning voids with ≥ 30% increase (geometric mean) in UACR from "run-in" period samples OR > 40 mg/g (geometric mean).

SECONDARY OUTCOMES:
Cardiovascular disease and mortality | Screening, (Low-risk: year 1, 2 and 3), (high-risk: week 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156)
  Comparison of composite fatal and non-fatal cardiovascular outcome (myocardial infarction, stroke, coronary artery bypass, coronary re-vascularisation, hospitalization for heart failure and cardiovascular death), and all-cause mortality during the study.
Retinopathy | Screening, (Low-risk: year 1, 2 and 3), (high-risk: week 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156)
  Comparison of incidence of retinopathy and frequency of laser treatment. Data collected from self-reported adverse events.
Change in albuminuria | Screening, (Low-risk: year 1, 2 and 3), (high-risk: week 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156)
  In addition to the categorical analysis of urinary albumin excretion, an analysis will be performed with changes in geometric mean albuminuria throughout the study period in all patients by assessing the slope of albuminuria changes and absolute changes from inclusion to end of trial
Microalbuminuria | Screening, (Low-risk: year 1, 2 and 3), (high-risk: week 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156)
  Development of microalbuminuria (UACR >30 mg/g) in at least one morn-ing void urine sample will be used as a secondary outcome instead of con-firmed microalbuminuria
Macroalbuminuria | Screening, (Low-risk: year 1, 2 and 3), (high-risk: week 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156)
  Development of macroalbuminuria (UACR >300 mg/g) in 2 out 3 first morning void urine samples)
Change in CKD class | Screening, (Low-risk: year 1, 2 and 3), (high-risk: week 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156)
  For patients with estimated GFR ≥ 60 at baseline, development of estimated GFR<60 ml/min/1.73m2. Estimated GFR will be measured from serum creatinine (standard-ized traceable method) on blood samples tested in local laboratories.
Slope of estimated GFR | Screening, (Low-risk: year 1, 2 and 3), (high-risk: week 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156)
  Change in estimated GFR (slope and absolute from baseline and from 3 month post-baseline to end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, Prof. MD, Study Chair — Steno Diabetes Center Copenhagen; Matias Trillini, MD, Principal Investigator — Istituto de Ricerche Farmacologiche Mario Negri; Alberto Ortiz, MD, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz; Christian Delles, MD, Principal Investigator — University of Glasgow; Gerjan Navis, MD, Principal Investigator — University Medical Center Groningen; Ivan Rychlik, MD, Principal Investigator — Univerzita Karlova v Praze; Joachim Beige, MD, Principal Investigator — Klinikum St. Georg gGmbH; Marina Noutsou, MD, Principal Investigator — Geniko Nosikomeico Athinas Ippokrateio, Hospital Diabetes Center; Peter Girman, MD, Principal Investigator — Institut Klinické a Experimentální Mediciny; Goce Spasovski, MD, Principal Investigator — Department of Nephrology, University of Skopje; Adriaan Kooy, MD, Principal Investigator — Diabetes Vascular Research Foundation Hoogeveen; Marjin Speeckaert, MD, Principal Investigator — University Ghent; Joline Beulens, MD, Principal Investigator — Stichting VUMC; Rüdiger Göke, MD, Principal Investigator — Diabetologen Hessen; Andreas Birkenfeld, MD, Principal Investigator — Universitätsklinikum Carl Gustav Carus, Technischen Universität Dresden
Locations (15):
- Universitair Ziekenhuis, Ghent, Belgium
- Czechia (2):
  - Institut Klinické a Experimentální Mediciny, Prague
  - Universita Karlova v Praze, Prague
- Steno Diabets Center Copenhagen, Gentofte Municipality, Denmark
- Germany (3):
  - Universitätsklinikum Carl Gustav Carus, Technischen Universität Dresden, Dresden
  - Diabetologen Hessen, Hessen
  - Klinikum St. Georg gGmbH, Leipzig
- Geniko Nosikomeico Athinas Ippokrateio, Hospital Diabetes Center, Athens, Greece
- Instituto de Ricerche Farmacologiche Mario Negri, Bergamo, Italy
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Diabetes Vascular Research Foundation, Hoogeveen
  - Stichting VUMC, Hoorn
- Department of Nephrology, University of Skopje, Skopje, North Macedonia
- Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz, Madrid, Spain
- University of Glasgow, Glasgow, United Kingdom

REFERENCES:
- [Derived] Rotbain Curovic V, Tofte N, Lindhardt M, Adamova K, Bakker SJL, Beige J, Beulens JWJ, Birkenfeld AL, Currie G, Delles C, Dimos I, Francova L, Frimodt-Moller M, Girman P, Goke R, Hansen TW, Havrdova T, Kooy A, Laverman GD, Mischak H, Navis G, Nijpels G, Noutsou M, Ortiz A, Parvanova A, Persson F, Petrie JR, Ruggenenti PL, Rutters F, Rychlik I, Siwy J, Spasovski G, Speeckaert M, Trillini M, Zurbig P, von der Leyen H, Rossing P; on the behalf of the PRIORITY Study Group. Presence of retinopathy and incident kidney and cardiovascular events in type 2 diabetes with normoalbuminuria - A post-hoc analysis of the PRIORITY randomized clinical trial. J Diabetes Complications. 2023 Apr;37(4):108433. doi: 10.1016/j.jdiacomp.2023.108433. Epub 2023 Feb 18. PMID 36841085
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- [Derived] Tofte N, Lindhardt M, Adamova K, Bakker SJL, Beige J, Beulens JWJ, Birkenfeld AL, Currie G, Delles C, Dimos I, Francova L, Frimodt-Moller M, Girman P, Goke R, Havrdova T, Heerspink HJL, Kooy A, Laverman GD, Mischak H, Navis G, Nijpels G, Noutsou M, Ortiz A, Parvanova A, Persson F, Petrie JR, Ruggenenti PL, Rutters F, Rychlik I, Siwy J, Spasovski G, Speeckaert M, Trillini M, Zurbig P, von der Leyen H, Rossing P; PRIORITY investigators. Early detection of diabetic kidney disease by urinary proteomics and subsequent intervention with spironolactone to delay progression (PRIORITY): a prospective observational study and embedded randomised placebo-controlled trial. Lancet Diabetes Endocrinol. 2020 Apr;8(4):301-312. doi: 10.1016/S2213-8587(20)30026-7. Epub 2020 Mar 2. PMID 32135136
- [Derived] Tofte N, Lindhardt M, Adamova K, Beige J, Beulens JWJ, Birkenfeld AL, Currie G, Delles C, Dimos I, Francova L, Frimodt-Moller M, Girman P, Goke R, Havrdova T, Kooy A, Mischak H, Navis G, Nijpels G, Noutsou M, Ortiz A, Parvanova A, Persson F, Ruggenenti PL, Rutters F, Rychlik I, Spasovski G, Speeckaert M, Trillini M, von der Leyen H, Rossing P. Characteristics of high- and low-risk individuals in the PRIORITY study: urinary proteomics and mineralocorticoid receptor antagonism for prevention of diabetic nephropathy in Type 2 diabetes. Diabet Med. 2018 Oct;35(10):1375-1382. doi: 10.1111/dme.13669. Epub 2018 Jun 6. PMID 29781558
- [Derived] Lindhardt M, Persson F, Currie G, Pontillo C, Beige J, Delles C, von der Leyen H, Mischak H, Navis G, Noutsou M, Ortiz A, Ruggenenti PL, Rychlik I, Spasovski G, Rossing P. Proteomic prediction and Renin angiotensin aldosterone system Inhibition prevention Of early diabetic nephRopathy in TYpe 2 diabetic patients with normoalbuminuria (PRIORITY): essential study design and rationale of a randomised clinical multicentre trial. BMJ Open. 2016 Mar 2;6(3):e010310. doi: 10.1136/bmjopen-2015-010310. PMID 26936907
- See also: Official study webpage — http://www.eu-priority.org
- See also: European Commission, The Seventh Framework Programme. — http://cordis.europa.eu/projects/rcn/101813_en.html

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT02040441/SAP_000.pdf
  • Study Protocol (2015-10-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT02040441/Prot_001.pdf